CLINICAL TRIAL: NCT00264849
Title: A Randomized, Open Label, Parallel-group, International, Multicenter Study Evaluating Persistency of Response to Omalizumab During 32 Weeks Treatment Given as Add on to Optimized Asthma Therapy in Adult and Adolescent Patients With Severe Persistent Allergic Asthma, Who Remain Inadequately Controlled Despite GINA (2004) Step 4 Therapy
Brief Title: Omalizumab in Adult and Adolescent Patients With Severe Persistent Allergic Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Genentech, Inc. (Industry); Tanox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIGE025A2425
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Results first posted 2011-07-25 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-04

CONDITIONS: Asthma
Keywords: Asthma; omalizumab; Severe persistent allergic asthma
MeSH Terms: conditions — Asthma | interventions — Omalizumab

ARMS (2):
- OAT + Omalizumab (Experimental): During the 8-week Run-in phase, asthma therapy was evaluated and optimized according to Global Initiative for Asthma (GINA) guidelines. During the treatment phase, participants continued to receive optimized asthma therapy (OAT), plus omalizumab add on therapy for 32 weeks, administered by subcutaneous injection once every 4 weeks. The dosage received was individualized based on body weight and serum IgE level.
  Interventions: Drug: Omalizumab; Other: Optimized asthma therapy
- Optimized Asthma Treatment (OAT) (Active Comparator): During the 8-week Run-in phase, asthma therapy was evaluated and optimized according to Global Initiative for Asthma (GINA) guidelines. In the treatment phase, participants continued to receive optimized asthma therapy (OAT) established during the run-in period of the study for 32 weeks.
  Interventions: Other: Optimized asthma therapy

INTERVENTIONS:
Drug: Omalizumab — Omalizumab administered by subcutaneous injection. The dosage received was individualized based on body weight and serum IgE level.
  Other Names: Xolair
  Arms: OAT + Omalizumab
Other: Optimized asthma therapy — Optimized asthma therapy (OAT) according to Global Initiative for Asthma (GINA) 2004 guidelines during the first 4 weeks of the run-in period of the study.

SUMMARY:
Omalizumab will be given as add-on treatment to optimized asthma therapy in patients with severe persistent asthma, who demonstrate inadequate asthma symptom control. Response to omalizumab over time will be assessed by physicians and patients evaluating the overall improvement in control of their asthma.

THIS STUDY IS NOT ENROLLING PATIENTS IN THE US.

ELIGIBILITY:
Inclusion Criteria:

Patients who met the following criteria were included:

* Males or females of any race, who were 12-75 years of age
* A body weight ≥ 20 kg and ≤ 150 kg and with a total serum IgE level ≥ 30 to ≤ 700 IU/ml
* A diagnosis of allergic asthma ≥ 1 year duration according to American Thoracic Society (ATS) criteria and at screening a history consistent with GINA (2204) step 3 or 4 clinical features
* A positive prick skin test (diameter of wheal >= 3 mm) to at least one perennial allergen documented within the past 2 years or taken at visit 1
* Increase in FEV1 ≥12% over baseline value within 30 minutes of taking 2 to 4 puffs (2-4x100µg) salbutamol (albuterol) or nebulized salbutamol up to 5mg
* An FEV1 ≥ 40 and ≤ 80% of the predicted normal value for the patient at randomization
* Receiving moderate to high dose inhaled corticosteroid ≥ 800 µg BDP or equivalent and a regular inhaled long acting B-2 agonists for at least 3 months prior to screening and > 1000 µg (BDP) and a LABA for at least 4 weeks during the run-in and at randomization
* Patients who have suffered multiple (i.e. at least two) independent documented severe asthma exacerbations while receiving high doses of ICS (≥ 800 µg BDP or equivalent) plus regular inhaled LABA
* Evidence of poor asthma control at screening (based on patient history) and for at least 4 weeks immediately prior to randomisation

Exclusion Criteria:

Patients who met the following criteria were excluded:

* Had received systemic corticosteroids for reasons other than asthma within 4 weeks of Visit 1
* A smoking history >10 pack years
* An active lung disease other than allergic asthma
* Elevated serum IgE levels for reasons other than allergy
* Patients with significant underlying medical conditions

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2005-11; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (17):
- Brussels, Belgium
- Montreal, Canada
- Hvidovre, Denmark
- Berlin, Germany
- Athens, Greece
- Budapest, Hungary
- Dublin, Ireland
- Haifa, Israel
- Roma, Italy
- Oslo, Norway
- Lodz, Poland
- Lisbon, Portugal
- Madrid, Spain
- Stockholm, Sweden
- Bern, Switzerland
- Bursa, Turkey (Türkiye)
- Nottingham, United Kingdom

REFERENCES:
- [Derived] Siergiejko Z, Swiebocka E, Smith N, Peckitt C, Leo J, Peachey G, Maykut R. Oral corticosteroid sparing with omalizumab in severe allergic (IgE-mediated) asthma patients. Curr Med Res Opin. 2011 Nov;27(11):2223-8. doi: 10.1185/03007995.2011.620950. Epub 2011 Sep 21. PMID 21933100

RESULTS

PARTICIPANT FLOW:
Groups:
- Optimized Asthma Treatment (OAT): During the 8-week Run-in phase, asthma therapy was evaluated and optimized according to Global Initiative for Asthma (GINA) guidelines. In the treatment phase, participants continued to receive optimized asthma therapy (OAT) established during the run-in period of the study for an additional 32 weeks.
Period: Overall Study
Arm/Group | OAT + Omalizumab | Optimized Asthma Treatment (OAT)
Started | 275 | 131
Completed | 253 | 106
Not Completed | 22 | 25
Not completed — Adverse Event | 7 | 2
Not completed — Withdrawal by Subject | 7 | 11
Not completed — Protocol Violation | 5 | 3
Not completed — Lack of Efficacy | 1 | 6
Not completed — Lost to Follow-up | 0 | 2
Not completed — Death | 0 | 1
Not completed — Administrative Problems | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OAT + Omalizumab | Optimized Asthma Treatment (OAT) | Total
Number analyzed (Participants) | 272 | 128 | 400
Age, Categorical [Count of Participants; unit: Participants] — All demographic data is described for the Modified ITT population. The modified ITT population includes all randomized patients with at least one post-baseline efficacy assessment
  Participants
    <=18 years | 5 | 0 | 5
    Between 18 and 65 years | 250 | 118 | 368
    >=65 years | 17 | 10 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (13.04) | 45.7 (12.57) | 45.7 (12.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 183 | 76 | 259
  Male | 89 | 52 | 141
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 266 | 125 | 391
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Persistency of Response and Non-response as Based on Investigator's Global Evaluation of Treatment Effectiveness (GETE)
Description: Persistency of response, based on GETE, was dichotomized into responders (excellent or good) and non-responders (moderate, poor or worsening). Persistent responders were patients who were responders at 16 weeks and still at 32 weeks. Persistent non-responders were patients who were non-responders at 16 weeks and still at 32 weeks. Patients were assessed for persistency of response if they were responders at Week 16 and had a second GETE obtained ≥ 4 weeks after the Week 16 assessment or discontinued prematurely for unsatisfactory therapeutic effect ≥ 4 weeks after the Week 16 assessment.
Time Frame: Weeks 16 and 32
Population: Modified Intent-to-Treat (mITT) was defined for efficacy analyses which included all randomized patients who had at least one post-baseline efficacy assessment.
Measure: Number; unit: participants
Arm/Group | OAT + Omalizumab | Optimized Asthma Treatment (OAT)
Number analyzed (Participants) | 272 | 128
participants
  Number of responders at Wk 16 | 190 | 29
  Participants available to assess persistency | 187 | 28
  Number of Persistent Responders at Weeks 16 and 32 | 171 | 18
  Number of non-responders at Week 16 | 71 | 64
  Participants to assess persistency of non respond | 71 | 63
  Number of Persistent Non-responders at Wks 16and32 | 44 | 57

2. Secondary Outcome: Number of Participants by Investigator's Global Evaluation of Treatment Effectiveness (GETE) Category at Week 16 and Week 32
Description: Number of participants with persistent response, based on the investigator's GETE, dichotomized to responders (excellent or good) and non-responders (moderate, poor or worsening) for patients receiving omalizumab as add on to optimal asthma therapy, assessed at week 16 and week 32. Persistency was defined as the proportion of responders at 16 weeks who were still responders at 32 weeks. GETE categories are excellent, good, moderate, poor, worsening, and missing as determined by the investigator.
Time Frame: Weeks 16 and 32
Population: Modified Intent-to-Treat (mITT)
Measure: Number; unit: participants
Arm/Group | OAT + Omalizumab | Optimized Asthma Treatment (OAT)
Number analyzed (Participants) | 272 | 128
participants
  Week 16: Excellent | 35 | 1
  Week 16: Good | 155 | 28
  Week 16: Moderate | 57 | 24
  Week 16: Poor | 13 | 34
  Week 16: Worsening | 1 | 6
  Week 16: Missing | 11 | 35
  Week 16: Responders (excellent and good) | 190 | 29
  Week 16: Non-responders (moderate, poor, worse) | 71 | 64
  Week 32: Excellent | 73 | 1
  Week 32: Good | 126 | 24
  Week 32: Moderate | 45 | 31
  Week 32: Poor | 13 | 39
  Week 32: Worsening | 2 | 9
  Week 32: Missing | 13 | 24
  Week 32: Responders (excellent and good) | 199 | 25
  Week 32: Non-responders (moderate, poor, worse) | 60 | 79
  Responder at both weeks (Weeks 16 and 32) | 171 | 18

3. Secondary Outcome: Percentage of Participants Who Were Responders at Both Week 16 and Week 32 Based on Investigator's GETE
Description: Responders were defined as excellent or good based on the investigator's Global Evaluation of Treatment Effectiveness (GETE) for patients receiving omalizumab as add on to optimal asthma therapy, assessed at week 16 and week 32.
Time Frame: Weeks 16 and 32
Population: Modified Intent-to-Treat (mITT)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OAT + Omalizumab | Optimized Asthma Treatment (OAT)
Number analyzed (Participants) | 272 | 128
percentage of participants | 62.9 [57.1 to 68.6] | 14.1 [8.0 to 20.1]

4. Secondary Outcome: Number of Participants by Patient's Global Evaluation of Treatment Effectiveness (GETE) Category at Week 16 and 32
Description: Number of participants with persistent response, based on the patient's GETE, dichotomized to responders (excellent or good) and non-responders (moderate, poor or worsening) for patients receiving omalizumab as add on to optimal asthma therapy, assessed at week 16 and week 32. Persistency was defined as the proportion of responders at 16 weeks who were still responders at 32 weeks. This is based on the patient's evaluation.
Time Frame: Weeks 16 and 32
Population: Modified Intent-to-Treat (mITT)
Measure: Number; unit: participants
Arm/Group | OAT + Omalizumab | Optimized Asthma Treatment (OAT)
Number analyzed (Participants) | 272 | 128
participants
  Week 16: Excellent | 54 | 4
  Week 16: Good | 139 | 29
  Week 16: Moderate | 53 | 23
  Week 16: Poor | 15 | 33
  Week 16: Worsening | 1 | 5
  Week 16: Missing | 10 | 34
  Week 16: Responders (excellent and good) | 193 | 33
  Week 16:Non-responders (moderate, poor, worsening) | 69 | 61
  Week 32: Excellent | 80 | 2
  Week 32: Good | 127 | 27
  Week 32: Moderate | 38 | 28
  Week 32: Poor | 12 | 38
  Week 32: Worsening | 2 | 8
  Week 32: Missing | 13 | 25
  Week 32: Responders (excellent and good) | 207 | 29
  Week 32: Non-responders (moderate, poor, worse) | 52 | 74

5. Secondary Outcome: Percentage of Participants Who Were Responders at Both Week 16 and Week 32 Based on Patient's GETE
Description: Responders were defined as excellent or good based on the patient's Global Evaluation of Treatment Effectiveness (GETE) for patients receiving omalizumab as add on to optimal asthma therapy, assessed at week 16 and week 32.
Time Frame: Weeks 16 and 32
Population: mITT population and patients who were assessed for persistency of response or non-response at Week 16 and had a GETE obtained >= 4 weeks after the Week 16 assessment or discontinued prematurely or unsatisfactory therapeutic effect >= 4 weeks after the Week 16 assessment. N=187/28 for OAT+Omalizumab/OAT for responders and N=71/63 for non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OAT + Omalizumab | Optimized Asthma Treatment (OAT)
Number analyzed (Participants) | 272 | 128
percentage of participants | 63.2 [57.5 to 69.0] | 15.6 [9.3 to 21.9]

6. Secondary Outcome: Lung Function Assessed by Forced Expiratory Volume for 1 Second (FEV1)
Description: Predicted FEV1 was calculated using the Crapo formula for data at Visit 6 (time of randomization), (MALES: Predicted FEV1 (L) = 0.0414*height - 0.0244*age -2.190 and Females: Predicted FEV1 (L) = 0.0342*height - 0.0255*age - 1.578, where height is in cm).
Time Frame: Weeks 16 and 32
Population: Modified Intent-to-Treat (mITT), for Week 16 N=258/106 for OAT+Omalizumab/OAT and for Week 32 N=266/121 for OAT+Omalizumab/OAT, respectively.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted FEV1
Arm/Group | OAT + Omalizumab | Optimized Asthma Treatment (OAT)
Number analyzed (Participants) | 272 | 128
percent predicted FEV1
  Week 16 | 68.4 [66.2 to 70.5] | 64.8 [61.8 to 67.8]
  Week 32 | 68.1 [65.8 to 70.5] | 63.7 [60.6 to 66.8]

7. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ) Overall Score at Weeks 16 and 32
Description: Asthma symptoms were evaluated by the Asthma Control Questionnaire (ACQ). The ACQ has six questions to be answered by the patient, each with a 7 point scale (0-good control, 6-poor control), and one question where the actual pre-bronchodilator FEV1 value expressed in % of predicted FEV1 was classified to scores from 0 (> 95% of predicted) to 6 (< 50% of predicted). The overall score is the average of the 7 questions; a minimum overall score of 0 = good control of asthma whereas a maximum overall score of 6 = poor control of asthma. A negative change in score indicates improvement in symptoms.
Time Frame: Baseline, Week 16, Week 32
Population: mITT with N counts as noted in the category description. To be included in this table patients must have a ACQ measurement for the specified timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OAT + Omalizumab | Optimized Asthma Treatment (OAT)
Number analyzed (Participants) | 272 | 128
units on a scale
  Week 16 (N=249,104) | -0.78 [-0.92 to -0.63] | -0.11 [-0.31 to 0.10]
  Week 32 (N=238,104) | -0.91 [-1.07 to -0.76] | -0.04 [-0.26 to 0.17]
  Last post-baseline (N=255,119) | -0.84 [-1.00 to -0.69] | 0.07 [-0.14 to 0.27]

8. Secondary Outcome: Number Participants With Clinically Significant Asthma Exacerbations by Category During the 32 Week Treatment Period
Description: A clinically significant exacerbation episode was defined as a worsening of asthma requiring treatment with rescue systemic (oral or IV) corticosteroids. The initiation of the rescue systemic corticosteroids marked the start of a clinically significant asthma exacerbation episode and cessation of the rescue systemic corticosteroids regimen marked the end of a clinically significant exacerbation episode. If an exacerbation episode was duplicated, overlapped by at least one day with another episode, or nested within another exacerbation episode, only one exacerbation was counted.
Time Frame: 32 Weeks
Population: mITT
Measure: Number; unit: participants
Arm/Group | OAT + Omalizumab | Optimized Asthma Treatment (OAT)
Number analyzed (Participants) | 272 | 128
participants
  0 asthma exacerbations | 183 | 64
  1 asthma exacerbation | 58 | 35
  2 asthma exacerbations | 18 | 17
  3 asthma exacerbations | 9 | 6
  >= 4 asthma exacerbations | 4 | 6

9. Secondary Outcome: Medical Resource Utilization: Number of Participants With Combined Hospital Admissions, Emergency Room Visits, and Other Outpatient Clinical Visits Due to an Asthma Exacerbation During the 32 Week Treatment Period
Description: A combined total of unscheduled visits due to asthma exacerbations was calculated for each patient as the total number of hospital admissions, ER visits and unscheduled outpatient clinical visits due to asthma exacerbation. Where more than one type of visit was required on a single day for an asthma exacerbation only the most serious type was included. Where there was more than one visit for a single asthma exacerbation but the visits occurred on different dates, then all were counted.
Time Frame: 32 Weeks
Population: Modified Intent-to-Treat (mITT)
Measure: Number; unit: participants
Arm/Group | OAT + Omalizumab | Optimized Asthma Treatment (OAT)
Number analyzed (Participants) | 272 | 128
participants
  0 combined visits/hospitalizations | 226 | 86
  1 combined visit/hospitalization | 26 | 12
  2 combined visits/hospitalizations | 10 | 17
  3 combined visits/hospitalizations | 4 | 8
  >= 4 combined visits/hospitalizations | 6 | 5
  Total number of combined visits/hospitalizations | 92 | 100

10. Secondary Outcome: Percent Change in Dose of Maintenance Systemic Steroids at Weeks 16 and 32
Description: For the subgroup of patients requiring maintenance oral (systemic) corticosteroids throughout the screening period the dose of oral steroid (expressed as prednisolone equivalent dose) at baseline, Week 16 and Week 32 was presented by treatment group, as well as the absolute and percent change from baseline to Weeks 16 and 32. It should be noted that the dose of oral steroid at Weeks 16 and 32 was the dose the patient was maintained on and not the dose to treat an exacerbation if one occurred at that time.
Time Frame: Weeks 16 and 32
Population: mITT patients with systemic steriods at baseline (defined as those patient who used systemic steroids throughout the entire run-in period from Visit 1 to Visit 6). N counts as noted in the category description.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | OAT + Omalizumab | Optimized Asthma Treatment (OAT)
Number analyzed (Participants) | 59 | 23
percent change
  Week 16 (N=56,19) | -20.1 (63.08) | 36.8 (212.03)
  Week 32 (N=59,23) | -45.0 (50.22) | 18.3 (85.13)

11. Secondary Outcome: Number of Participants by Type of Dose Change of Maintenance Systemic Steroids at Weeks 16 and 32
Description: The type of change for the dose of maintenance systemic steroids could be presented as removal (no more maintenance systemic steroids used), decreased, or maintained.
Time Frame: Weeks 16 and 32
Population: mITT patients with systemic steroids at baseline (defined as those patient who used systemic steroids throughout the entire run-in period from Visit 1 to Visit 6).
Measure: Number; unit: participants
Arm/Group | OAT + Omalizumab | Optimized Asthma Treatment (OAT)
Number analyzed (Participants) | 59 | 23
participants
  Week 16 - Removed systemic steroids (N=56,19) | 10 | 2
  Week 16 - Decreased systemic steroids (N=56,19) | 14 | 2
  Week 16 - Maintained systemic steroids (N=56,19) | 32 | 15
  Week 32 - Removed systemic steroids | 19 | 3
  Week 32 - Decreased systemic steroids | 18 | 4
  Week 32 - Maintained systemic steroids | 22 | 16

12. Secondary Outcome: Change From Baseline in Asthma Quality of Life Questionnaire (AQLQ) Overall Score by Visit
Description: There are 32 questions in the AQLQ and they are in 4 domains (symptoms, activity limitation, emotional function and environmental exposure). Each question was answered on a 7 point scale (1-totally limited/problems all the time, 7-not at all limited/no problems). The overall AQLQ score is the mean of all 32 responses, and the individual domain scores are the means of the items in those domains (a minimum domain / overall score of 1 = Severely impaired whereas a maximum domain / overall score of 7 = not impaired at all). A positive change from baseline score indicates improvement.
Time Frame: Baseline, Week 15, Week 31
Population: mITT at Week 15 for OAT + Omalizumab is 214 patients and for OAT is 92 patients; at Week 31 for OAT + Omalizumab is 224 patients and for OAT is 97 patients except as noted in the category description. To be included in this table patients must have a AQLQ measurement for the specified timepoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OAT + Omalizumab | Optimized Asthma Treatment (OAT)
Number analyzed (Participants) | 272 | 128
units on a scale
  Overall Score: Week 15 | 0.90 [0.73 to 1.07] | 0.03 [-0.20 to 0.27]
  Overall Score: Week 31 | 1.06 [0.88 to 1.24] | -0.07 [-0.31 to 0.17]
  Symptom Score: Week 15 | 0.89 [0.70 to 1.09] | -0.05 [-0.31 to 0.22]
  Symptom Score: Week 31 | 1.07 [0.88 to 1.27] | -0.07 [-0.34 to 0.19]
  Activities Score: Week 15 | 0.87 [0.70 to 1.04] | 0.03 [-0.20 to 0.26]
  Activities Score: Week 31 | 1.08 [0.91 to 1.26] | -0.07 [-0.31 to 0.17]
  Emotions Score: Week 15 | 0.98 [0.78 to 1.18] | 0.20 [-0.07 to 0.48]
  Emotions Score: Week 31 | 1.08 [0.88 to 1.28] | -0.07 [-0.34 to 0.19]
  Enironmental Exposure Score: Week 15 (N=213,91) | 0.84 [0.66 to 1.02] | 0.10 [-0.15 to 0.34]
  Enironmental Exposure Score: Week 31(N=223,96) | 0.91 [0.71 to 1.11] | -0.01 [-0.29 to 0.26]

13. Secondary Outcome: Change From Baseline in EuroQual 5-Dimension Health Status Questionnaire (EQ-5D) Index Score and Health State Assessment on Scale From 0 to 100 at Weeks 15 and 31
Description: The utility-based EQ-5D questionnaire is in two parts and provides a generic measure of health for clinical and economic appraisal. The first "health state classification" part has 5 questions each with 3 categories (no problem, moderate problem, severe problems). The second "visual analogue scale" was measured from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline, Week 15, Week 31
Population: Modified Intent-to-Treat with N count as noted in category description.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OAT + Omalizumab | Optimized Asthma Treatment (OAT)
Number analyzed (Participants) | 272 | 128
units on a scale
  EQ-5D Utility Index Score: Week 15 (N=212,90) | 0.071 [0.038 to 0.105] | 0.002 [-0.044 to 0.049]
  EQ-5D Utility Index Score: Week 31 (N=194,81) | 0.091 [0.051 to 0.132] | 0.064 [0.008 to 0.121]
  Health State Assessment: Week 15 (N=211,89) | 8.2 [4.7 to 11.8] | -0.4 [-5.4 to 4.6]
  Health State Assessment: Week 31 (N=194,80) | 9.3 [5.2 to 13.4] | -2.8 [-8.5 to 3.0]

14. Secondary Outcome: Changes From Baseline to Week 31 in the Percent Overall Work Impairment Due to Asthma Problems
Description: The Work Productivity and Activity Impairment-Allergic Asthma (WPAI-AA) questionnaire measures time missed from work, impairment of work and regular activities within the last 7 days. Questionnaires were administered via phone 1 week prior to the study visit. Outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity. Overall work impairment due to asthma problems is derived from the proportion of hours missed from work due to asthma and the degree to which asthma problems affected productivity while working.
Time Frame: Baseline and Week 31
Population: Modified Intent-to-Treat. Only patients only who worked and with values at both baseline and Week 31 visit were included. Sensitivity analysis excluded questionnaires which were answered after the clinic visit.
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | OAT + Omalizumab | Optimized Asthma Treatment (OAT)
Number analyzed (Participants) | 78 | 32
percent impairment
  Baseline | 41.3 (26.19) | 39.4 (24.91)
  Week 31 | 20.5 (24.28) | 40.3 (27.97)
  Change from baseline at Week 31 | -20.8 (26.38) | 0.8 (30.34)

ADVERSE EVENTS:
Arm/Group | OAT + Omalizumab | Optimized Asthma Treatment (OAT)
Serious Adverse Events (participants affected / at risk) | 29/274 | 17/128
Other Adverse Events (participants affected / at risk) | 140/274 | 65/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OAT + Omalizumab (N=274) | Optimized Asthma Treatment (OAT) (N=128)
Cardiac arrest (Cardiac disorders) | 1 | 0
Goitre (Endocrine disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Polyp (General disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Orchitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 15 | 14
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OAT + Omalizumab (N=274) | Optimized Asthma Treatment (OAT) (N=128)
Bronchitis (Infections and infestations) | 13 | 7
Influenza (Infections and infestations) | 18 | 4
Lower respiratory tract infection (Infections and infestations) | 16 | 8
Nasopharyngitis (Infections and infestations) | 38 | 9
Sinusitis (Infections and infestations) | 10 | 7
Upper respiratory tract infection (Infections and infestations) | 17 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 0
Headache (Nervous system disorders) | 33 | 9
Asthma (Respiratory, thoracic and mediastinal disorders) | 82 | 51
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.